CLINICAL TRIAL: NCT02877524
Title: Trial to Study Intubation Rates of Non-invasive Ventilation Using Pressure Support Ventilation (PSV) Versus Adaptive Support Ventilation (ASV) Mode in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: PSV vs ASV for
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Department of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NK/2609/DM/105
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Invasive Mechanical Ventilation; Adaptive Support Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive support ventilation (Experimental): Adaptive support ventilation during NIV for acute exacerbation of COPD
  Interventions: Other: Adaptive support ventilation
- Pressure support ventilation (Active Comparator): Pressure support ventilation during NIV for acute exacerbation of COPD
  Interventions: Other: Pressure support ventilation

INTERVENTIONS:
Other: Adaptive support ventilation — ASV during NIV
  Other Names: ASV
  Arms: Adaptive support ventilation
Other: Pressure support ventilation — PSV during NIV
  Other Names: PSV
  Arms: Pressure support ventilation

SUMMARY:
The clinical course of chronic obstructive pulmonary disease (COPD) is associated with recurrent episodes of exacerbation that results in respiratory failure. The treatment of respiratory failure is supportive and involves inhalation bronchodilators along with systemic steroids. In few cases the management of acute respiratory failure requires positive pressure ventilation (non-invasive or invasive). The use of NIV in acute exacerbation of COPD has resulted in significant reduction in morbidity and mortality. Although pressure support ventilation (PSV) allows the patient to influence the breathing pattern, ventilator-cycling criteria may worsen the patient-ventilator interaction, and severe asynchronies occur in up to 43% of patients undergoing NIV for ARF. Adaptive support ventilation (ASV) is a newer mode of ventilation that incorporates feedback mechanisms and thus provides a stable minute ventilation. We hypothesize that the use of ASV as a mode during ventilation using NIV in patients with acute exacerbation of COPD may result in reducing the duration of ventilatory support, need for intubation, and duration of intensive care unit (ICU) and hospital length of stay, when compared with PSV mode of NIV ventilation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common respiratory disease, which is characterized by airflow limitation. It affects more than 3.49 per cent of adults >35 year and is associated with high morbidity and mortality. The national burden of chronic bronchitis is estimated at 14.84 million.

The clinical course of COPD is punctuated by acute exacerbations, which can lead to hypercapnic respiratory failure. The development of respiratory failure is associated with high morbidity and mortality, and significant healthcare costs. The requirement of ventilatory support also portends a reduced survival in this group of patients.

The introduction of non-invasive ventilation (NIV) has resulted in a paradigm shift in the management of patients with acute exacerbation of COPD. First, reported in 1989, by Meduri et all, the successful application of NIV via full-face mask in 10 patients, and the avoidance of intubation in 8 of them (4 of 6 with COPD, 2 of 2 with congestive heart failure, and 2 of 2 with pneumonia), demonstrated the efficacy of NIV in the management of acute exacerbation of COPD. This new modality was successful in avoiding of many of the complications associated with invasive mechanical ventilation.

Traditionally, NIV is instituted with the pressure support mode of ventilation. Wherein, the inspiratory pressure was initiated at 6-8 cm of water and expiratory pressure was set at 3-4 cm. The difference between the two pressures provided the ventilatory support. These pressures were then titrated based on patient clinical improvement by the physician.

Adaptive support ventilation (ASV) is one of the newer modes of ventilation, described by Tehrani et al in 1991 and was designed to minimise the work of breathing, mimic natural breathing and stimulate breathing and reduce weaning time. It is a closed loop system, which incorporates various feedback mechanisms into its algorithm. The operator inputs patients weight, from that the ventilator calculates required minute alveolar ventilation assuming normal dead space fraction. Then an optimal frequency is calculated based on Otis equation. The target tidal volume is calculated by MV/f. The inspiratory pressure within a breath is controlled to achieve a constant value and between the breaths the inspiratory pressure is adjusted to achieve a target tidal volume. It aims to provide a target minute ventilation by adjusting automatically the delivered pressure and respiratory rate while keeping the work of breathing to a minimum by the patient.

Due to its ability to reduce the work of breathing and meet the flow requirement of the patient by adjusting both the flow and respiratory rate depending on the respiratory mechanics, the use of ASV as a mode of ventilation during NIV may improve patient-ventilator synchrony. A study comparing ASV versus pressure support ventilation in intubated patients with acute exacerbation of COPD demonstrated that the use of ASV mode was associated with shorter weaning times with similar weaning success rates. However, a study comparing the use of ASV mode versus PSV mode during non-invasive ventilation has not been done previously. Patient-ventilator synchronization is critical for reducing the work of breathing and for successful NIV. Although PSV allows the patient to influence the breathing pattern, ventilator-cycling criteria may worsen the patient-ventilator interaction, and severe asynchronies occur in up to 43% of patients undergoing NIV for ARF. We hypothesize that the use of ASV as a mode during ventilation using NIV in patients with acute exacerbation of COPD may result in reducing the duration of ventilatory support, need for intubation, and duration of intensive care unit (ICU) and hospital length of stay, when compared with PSV mode of NIV ventilation.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with acute exacerbation of COPD will be assessed for inclusion in the current study. The diagnosis of acute exacerbation of COPD will be made based on following criteria:

1. an acute sustained worsening of any of the patient's respiratory symptoms (cough, sputum quantity and/or character, dyspnea) that is beyond normal day today variation and leads to a change in medication
2. arterial blood gas analysis showing a PaCO2>45 mm of Hg with either pH <7.35 ≥7.26 or respiratory rate >30/minute
3. exclusion of other causes of acute breathlessness such as acute heart failure, pulmonary embolism, pneumonia, and pneumothorax.

Exclusion Criteria:

Patients with any one of the following criteria will be excluded from the current study:

1. non-COPD acute hyper-capneic respiratory failure.
2. hypotension (systolic blood pressure<90mmHg),
3. severe encephalopathy (Glasgow coma scale score < 8),
4. upper gastrointestinal bleeding
5. inability to protect the airway and clear respiratory secretions, or abnormalities that preclude proper fit of the interface (agitated or uncooperative patient, facial trauma or burns, facial surgery, or facial anatomical abnormality).
6. patients who are on home NIV.
7. failure to give consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of NIV success | 28 days after discharge
  To assess the difference in the rate of NIV success using either PSV or ASV mode of ventilation

SECONDARY OUTCOMES:
Patient comfort | 28 days after discharge
  Assess patient comfort using VAS score
Duration of mechanical ventilation | 28 days after discharge
  Duration of mechanical ventilation (both non-invasive and invasive)
Time to weaning | 28 days after discharge
  Total time to wean from positive airway pressure ventilation
ICU and hospital length of stay | 28 days after discharge
  Total duration of hospital and intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, Study Director — PGIMER,Chandigarh
Locations (1):
- Respiratory ICU, Post Graduate Institue of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sehgal IS, Kalpakam H, Dhooria S, Aggarwal AN, Prasad KT, Agarwal R. A Randomized Controlled Trial of Noninvasive Ventilation with Pressure Support Ventilation and Adaptive Support Ventilation in Acute Exacerbation of COPD: A Feasibility Study. COPD. 2019 Apr;16(2):168-173. doi: 10.1080/15412555.2019.1620716. Epub 2019 Jun 4. PMID 31161812